CLINICAL TRIAL: NCT02222311
Title: Influence of Vitamin D Deficiency on the Development of Autism
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0038-14-HYMC
Record Dates: First submitted 2014-08-11; First posted 2014-08-21 (Estimated); Last update posted 2014-08-21 (Estimated); Status verified 2014-08

CONDITIONS: Autism
MeSH Terms: conditions — Autistic Disorder | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Autistic Children: Children diagnosed with autism spectrum disorder according to the criteria of the Diagnostic Statistical Manual-V will have blood samples taken for laboratory analysis.
  Interventions: Other: Blood Samples
- Healthy Children: Children with no developmental or physical diseases will have blood samples taken for laboratory analysis.
  Interventions: Other: Blood Samples
- Children with Attention Deficit Disorder: Blood samples from children with Attention Deficit Disorder will be measured for Vitamin D and oxidative stress markers.
  Interventions: Other: Blood Samples

INTERVENTIONS:
Other: Blood Samples

SUMMARY:
The investigators wish to study the effect of Vitamin D on the development of autism in children. The investigators will also investigate the environmental and genetic influences on the level of Vitamin D in children with autism.

ELIGIBILITY:
Inclusion Criteria:

* Autistic children
* Healthy children
* Children with ADD

Exclusion Criteria:

* All others

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children with autism who have presented to the Child Development Institute at the Hillel Yaffe Medical Center and from pediatric neurology community clinics. The control groups include healthy age-matched children and children with Attention Deficit Disorder (ADD) who have presented to the Child Development Institute at the Hillel Yaffe Medical Center and from pediatric neurology community clinics.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2014-11; Primary Completion 2017-11 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Level of Vitamin D | One day
  Blood samples of patients with and without autism with be taken and the level of vitamin D in their serum will be determined (international units).

SECONDARY OUTCOMES:
Effect of environment on Vitamin D level | One week
  All participant blood samples will be measured for levels of oxidative stress markers and antioxidants.

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel